CLINICAL TRIAL: NCT05785611
Title: A Phase 3 Randomized, Placebo-controlled, Double-blind, Parallel-group Program to Evaluate Efficacy and Safety of Filgotinib in Adult Subjects With Active Axial Spondyloarthritis
Brief Title: A Study Evaluating the Effect of Filgotinib in Participants With Active Axial Spondyloarthritis
Acronym: OLINGUITO
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alfasigma S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GLPG0634-CL-336; 2022-501354-10-01 (EU CTIS Number)
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Axial Spondyloarthritis
Keywords: chronic inflammatory disease
MeSH Terms: conditions — Axial Spondyloarthritis | interventions — GLPG0634

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radiographic Part (Study A) Filgotinib (Experimental): Participants will receive filgotinib 200 mg or placebo to match filgotinib. Participants will receive blinded treatment until Week 16. After that participants with an age under 65 and without certain health risks will enter open label period and will receive filgotinib 200 mg until Week 52. Participants reaching an Ankylosing Spondylitis Disease Activity Score (ASDAS) <2.1 at weeks 40 and 52, will enter dose de-escalation phase and will be randomized to filgotinib 200 or 100 mg until Week 104. Participants, with an age of 65 or above or with certain health risks, will enter open label period until Week 104 and will receive 100 or 200 mg filgotinib a day, depending on their axSpA symptoms. The maximum duration of treatment period will be up to Week 104.
  Where applicable, participants will be able to enter an open-label extension period until week 234.
  Interventions: Drug: Filgotinib; Drug: Placebo
- Non-radiographic Part (Study B) Filgotinib (Experimental): Participants will receive filgotinib 200 mg or placebo to match filgotinib. Participants will receive blinded treatment until Week 16. After that participants with an age under 65 and without certain health risks will enter open label period and will receive filgotinib 200 mg until Week 52. Participants reaching an ASDAS <2.1 at weeks 40 and 52, will enter dose de-escalation phase and will be randomized to filgotinib 200 or 100 mg until Week 104. Participants, with an age of 65 or above or with certain health risks, will enter open label period until Week 104 and will receive 100 or 200 mg filgotinib a day, depending on their axSpA symptoms. The maximum duration of treatment period will be up to Week 104.
  Where applicable, participants will be able to enter an open-label extension period until week 234.
  Interventions: Drug: Filgotinib; Drug: Placebo

INTERVENTIONS:
Drug: Filgotinib — Tablets administered orally once daily
  Other Names: GS-6034; GLPG0634
Drug: Placebo — Tablets administered orally once daily

SUMMARY:
This study is comparing 200 milligrams (mg) of filgotinib a day with a placebo to see if filgotinib helps to treat Axial Spondyloarthritis (axSpA) and is safe to use. The study will also be comparing 200 mg with 100 mg filgotinib a day to see if the lower dose also helps to treat axSpA.

ELIGIBILITY:
Key Inclusion Criteria:

* Have an established diagnosis of axSpA by a rheumatologist (or other specialist with expertise in diagnosing axSpA).
* Study A (r-axSpA): Meet Assessment of SpondyloArthritis International Society (ASAS) classification criteria with radiographic sacroiliitis on X-ray as follows:

  1. History of back pain >=12 weeks and age at onset of back pain <45 years, AND
  2. Have radiographic bilateral grade 2-4 sacroiliitis or unilateral grade 3-4 sacroiliitis, based on New York grading system, confirmed by central reading, AND,
  3. >=1 spondyloarthritis (SpA) feature.
* Study B (nr- axSpA): Meet ASAS classification criteria without radiographic sacroiliitis on X-ray as follows:

  1. History of back pain >= 12 weeks and age at onset of back pain <45 years, AND
  2. No radiographic bilateral grade 2-4 sacroiliitis or unilateral grade 3-4 sacroiliitis, AND,
  3. Presence of sacroiliitis on MRI (based on central reading) and at least 1 SpA feature or when positive for human leukocyte antigen (HLA)-B27: having at least 2 SpA features, AND
  4. Have objective signs of inflammation, by sacroiliitis on MRI or elevated CRP.
* Have active axSpA at screening and Day 1 defined by:

  * Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) >=4 (numeric rating scale [NRS] 0-10), AND
  * Spinal pain score >=4 (0-10 NRS) (based on BASDAI question 2),
* Have a history of inadequate response to >=2 NSAIDs at the maximum dose of NSAIDs used in axSpA for >=2 weeks each (a total duration of NSAID trial >=4 weeks) or intolerance to >=2 NSAIDs for the treatment of axSpA.
* Participants who are biologic disease-modifying antirheumatic drug (BDMARD)(s) experienced; defined as below.

  * Participants designated as bDMARD(s)-inadequate responder(IR) must have received not more than 2 bDMARD(s), that was/were administered in accordance with its/their labeling and discontinued due to:

    * Non-response (primary or secondary) after a minimum treatment of 12 weeks, and /or
    * Intolerance (defined as having experienced an adverse reaction [e.g. an infusion/injection reaction, an infection, a laboratory test change, etc] irrespective of treatment duration)
  * Participants designated as bDMARD(s) non-IR have previously received bDMARD(s) and have discontinued these due to other reasons than non-response or intolerance (e.g. economic reasons, treatment as part of a clinical study, other, or unknown).
* If continuing conventional synthetic disease-modifying antirheumatic drugs (csDMARDs) during the study, participants are permitted to use only a maximum of 2 csDMARDs and must have been on this treatment for >=12 weeks prior to screening, with a stable dose and route of administration (defined as no change in prescription) for >4 weeks prior to Day 1.
* For participants aged 65 years or above on the date of signing the informed consent form (ICF), the investigator should carefully consider if participation is in the best interest of the participant.

Key Exclusion Criteria:

* Prior exposure to a Janus kinase inhibitor, investigational or approved, at any time, including filgotinib.
* Use of any opioid analgesic at average daily doses >30 mg/day of morphine (or equivalent) or use of unstable doses of any opioid analgesic <=2 weeks prior to Day 1.
* Use of any of the following systemic immunomodulating therapies <= 4 weeks prior to Day 1, including, but not limited to: 6-mercaptopurine, azathioprine, cyclosporine or other calcineurin inhibitors (e.g. sirolimus, tacrolimus), methotrexate if being discontinued, mycophenolate, antimalarials (e.g. hydroxychloroquine, chloroquine) if being discontinued, or sulfasalazine if being discontinued.
* Complete spinal ankylosis defined as the presence of consecutive bridging syndesmophytes in >=5 segments on the lateral radiograph (assessed by the central reader).
* Have undergone surgical treatments for peripheral manifestation of axSpA, including synovectomy or arthroplasty, or major surgery (requiring regional block or general anesthesia) <=12 weeks prior to Day 1 or planned major surgery during the study.
* Have a diagnosis of any generalized musculoskeletal disorder, e.g. generalized osteoarthritis, or systemic inflammatory condition other than axSpA.
* Have active Crohn's disease (CD) or active ulcerative colitis (UC). Note: participants may be enrolled if they have had a history of inflammatory bowel disease (IBD), including CD and UC, but have had no exacerbation within 6 months prior to Day 1, and, if currently on treatment, must be on stable treatment for >=6 months prior to Day 1 and this treatment should be allowed per protocol.
* Active autoimmune disease that would interfere with assessment of study parameters or increase risk to the participant by participating in the study (e.g. uncontrolled uveitis, uncontrolled thyroiditis, transverse myelitis, current peptic ulcer disease or prior history of severe diverticulitis [i.e. requiring hospitalization] or previous gastrointestinal perforation), per judgment of investigator,
* History of opportunistic infection, or immunodeficiency syndrome, which would put the participant at risk, as per investigator judgment,
* Active infection that is clinically significant, as per judgment of the investigator, or history of a serious infection (requiring hospitalization or systemic antibiotics) within 12 weeks prior to screening.
* Participant has a history of malignancy or myelo- or lymphoproliferative disorder, including non-melanoma skin cancer (NMSC), excised and curatively treated non-metastatic basal cell carcinoma, squamous cell carcinoma of the skin, or in situ uterine cervical carcinoma within the past 5 years prior to screening.
* Participant has any other condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (e.g. compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments. For participants at increased risk of major cardiovascular problems (such as heart attack or stroke), those who smoke or have done so for a long time in the past (>10 pack-years) and those at increased risk of cancer, the investigator should carefully consider if participation is in the best interest of the participant.
* Contraindication to magnetic resonance imaging (MRI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving SpondyloArthritis International Society 40% improvement (ASAS40) Response (Yes/No) at Week 16 | Week 16

SECONDARY OUTCOMES:
Change from baseline in Ankylosing Spondylitis DiseaseActivity Score with C-reactive protein (ASDASCRP) at Week 16 | Week 16
Change from baseline in Spondyloarthritis Research Consortium of Canada (SPARCC) Magnetic Resonance Imaging (MRI) Score of Sacroiliac Joints (SIJs) at Week 16 | Week 16
Change from baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) at Week 16 | Week 16
Change from baseline in Ankylosing Spondylitis Quality of Life (ASQoL) at Week 16 | Week 16
Change from baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI) (linear score) at Week 16 | Week 16
Number of Participants With Treatment-Emergent Adverse Events (TEAEs), TE Serious Adverse Events, and TEAEs Leading to Treatment Discontinuation at Week 16 | Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Alfasigma Study Director, Study Director — Alfasigma S.p.A.
Locations (123):
- Belgium (5):
  - Cliniques Universitaires de Bruxelles Hopital Erasme, Brussels
  - ReumaClinic, Genk
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
  - CHU Helora, Mons
- Bulgaria (16):
  - Medical Center Rodopimed, Kardzhali
  - MC Medconsult Pleven, Pleven
  - UMHAT Plovdiv AD, Plovdiv
  - UMHAT Eurohospital Plovdiv, Plovdiv
  - Medical Center UNIMED EOOD, Plovdiv
  - Medical Center Teodora, Rousse
  - Medical Center 1 Sevlievo, Sevlievo
  - DCC Ascendent EOOD, Sofia
  - UMHAT Sofiamed OOD, Sofia
  - Dcc Focus 5 Meoh Ood, Sofia
  - Dcc Focus 5 Meoh, Sofia
  - DCC XVII-Sofia EOOD, Sofia
  - Medical Center Hera, Sofia
  - Medical Center N I PIROGOV, Sofia
  - Military Medical Academy MHAT, Sofia
  - UMHAT Stoyan Kirkovich AD, Stara Zagora
- Czechia (14):
  - Lekarna U Revmatologickeho, Prague, Nove Mesto
  - Fakultni nemocnice u sv Anny, Interni klinika, Brno
  - Revmaclinic s r o, Brno
  - Lekarna BENU, Brno
  - Revmatologie s r o, Brno
  - CCR Ostrava, Ostrava
  - Vesalion Revma ambulance, Ostrava
  - Artroscan s r o, Ostrava
  - ARTHROHELP s r o, Pardubice
  - CCR Czech a s, Pardubice
  - MUDR. Zuzana URBANOVA Revmatologie, Prague
  - Fakultni nemocnice Motol, Prague
  - Medical Plus Sro, Uherské Hradiště
  - PV Medical Services, Zlín
- Estonia (2):
  - Clinical Research Centre, Tartu
  - Meditrials OU, Tartu
- France (5):
  - APHP Hopital Ambroise Pare, Boulogne-Billancourt
  - Hopital Edouard Herriot, Lyon
  - CHR d'Orleans, Orléans
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hopital Charles Nicolle, Rouen
- Germany (5):
  - Charite Medizinische Klinik I, Berlin
  - Hamburger Rheuma II, Hamburg
  - Rheumazentrum Ruhrgebiet, Herne
  - Klinische Forschung im med, Planegg
  - Universitatsklinikum Wurzburg, Würzburg
- Hungary (5):
  - Revita Rheumatologiai Kft, Budapest
  - University of Debrecen, Debrecen
  - Reumatologiai es Immunologiai, Pécs
  - Vita Verum Medical, Székesfehérvár
  - Obudai Egeszsegugyi Centrum, Zalaegerszeg
- Italy (6):
  - Istituto Ortopedico Rizzoli, Bologna
  - Azienda Ospedaliera Universitaria Luigi Vanvitelli, Napoli
  - Policlinico Paolo Giaccone, Palermo
  - Policlinico Uni Campus Bio-Med, Rome
  - Policlinico Universitario Agostino Gemelli, Rome
  - Ospedale SM Misericordia, Udine
- Lithuania (4):
  - Kaunas Hospital of LUHSCP, Kaunas
  - Kaunas City Polyclinic, Kaunas
  - Klaipeda University Hospital, Public Institution, Klaipėda
  - Vilnius UH Santariskiu Clinics, Vilnius
- Netherlands (2):
  - Medisch Spectrum Twente, Enschede
  - Medisch Centrum Leeuwarden, Leeuwarden
- Philippines (8):
  - Ilocos Training and Regional Medical Center, San Fernando City, La Union
  - Ospital Ng Makati, Makati City, National Capital Region
  - Lipa Medix Medical Center, Lipa City
  - Mary Mediatrix Medical Center, Lipa City
  - Medical Center Manila, Manila
  - The Medical City Clark, Mabalacat, Pampanga
  - St. Luke's Medical Center, Quezon City
  - Far Eastern University - Dr. Nicanor Reyes Medical Foundation, Quezon City
- Poland (18):
  - ZDROWIE Osteo Medic, Bialystok
  - Centrum Kliniczno Badawcze, Elblag
  - Silmedic sp. z o. o, Katowice
  - Reumed Spolka z o o, Lubin
  - KO-MED Centra Kliniczne, Lublin
  - Twoja Przychodnia NCM, Nowa Sól
  - ETYKA Osrodek Badan Klinicznyc, Olsztyn
  - TPO Centrum Medyczne, Opole
  - Solumed Medical Center, Poznan
  - AI Centrum Medyczne, Poznan
  - Twoja Przychodnia PCM, Poznan
  - KO-MED Centra Kliniczne, Staszów
  - MICS Medical Center Torun, Torun
  - MICS Centrum Medyczne, Warsaw
  - Instytut Reumatologii im. Eleonory Reicher, Warsaw
  - ETG Warszawa, Warsaw
  - Klinika Reuma Park, Warsaw
  - FutureMeds Wroclaw, Wroclaw
- Romania (9):
  - Sj de Urgenta Bacau, Bacau
  - S.C Centrul Medical de Diagnostic si Tratament Ambulator Neomed S.R.L, Brasov
  - SC Delta Health Care SRL, Bucharest
  - Spitalul Clinic Judetean de Urgenta, Cluj-Napoca
  - Aqua Med Consulting SRL, Constanța
  - SC Medisof Diagnostic SRL, Craiova
  - Centrul Medical Unirea SRL, Iași
  - Sc Medaudio Optica Srl, Râmnicu Vâlcea
  - S.C Centrul Medical Unirea SR, Târgu Mureş
- South Africa (4):
  - Clinresco Centres Pty Ltd,, Kempton Park
  - Arthritis Clinical Trial Centre, Pinelands
  - Emmed Research, Pretoria
  - Winelands Medical Research Centre, Stellenbosch
- South Korea (6):
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
- Spain (9):
  - Hospital Marina Baixa, Alicante
  - UH Parc Tauli, Barcelona
  - Hospital Universitario Basurto, Bilbao
  - HU Reina Sofia, Córdoba
  - Hospital Universitario La Paz, Madrid
  - HU Marques de Valdecilla, Santander
  - Clinica GAIAS Santiago, Santiago de Compostela
  - HU Virgen Macarena, Seville
  - UH Virgen de Valme, Seville
- Taiwan (3):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taipei Medical University Hospital, Taipei
- United Kingdom (2):
  - Royal United Hospital Bath NHS Foundation Trust, Bath
  - Norfolk & Norwich University Hospital, Norwich

IPD SHARING:
Plan to Share IPD: No